CLINICAL TRIAL: NCT01678560
Title: Remote Monitoring in Obstructive Sleep Apnea Management in Military Veterans
Brief Title: Remote Monitoring in Obstructive Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was halted due to the difficulties in recruiting.
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 01648
Record Dates: First submitted 2012-08-30; First posted 2012-09-05 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea PAP adherence efficacy economics
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Monitoring every 3 months by face-to-face visits:These patients will be monitored on a 3-month, 6-month, 9-month and 12-month intervals with scheduling face-to-face visits. Adherence and efficacy data will only be assessed by the clinician at these intervals.
  Interventions: Device: Monitoring every 3 months by face-to-face visits
- Wireless Care (Active Comparator): Frequent remote monitoring:These patients will be monitored using wireless modems as the method to obtain adherence and efficacy data.
  Interventions: Device: Frequent remote monitoring

INTERVENTIONS:
Device: Monitoring every 3 months by face-to-face visits — These patients will be monitored on a 3-month, 6-month, 9-month and 12-month intervals with scheduling face-to-face visits. Adherence and efficacy data will only be assessed by the clinician at these intervals.
  Arms: Usual Care
Device: Frequent remote monitoring — These patients will be monitored using wireless modems as the method to obtain adherence and efficacy and follow-up phone calls
  Arms: Wireless Care

SUMMARY:
Obstructive sleep apnea (OSA) among Veterans is a condition that imparts a great burden to the patient in terms of serious co-morbidities and results in a great cost to the VA Health Care System to treat the co-morbidities, which include heart disease, stroke and neuropsychiatric disorders. Positive airway pressure (PAP) is used to treat sleep apnea and studies have shown a poor adherence to treatment. The investigators hypothesize that using wireless technology will lead to early detection of problems of treatment use and will translate into early remedial action which will improve the use and effectiveness of treatment. The investigators will compare two methods. Usual care involves downloading data from PAP machines at designated 3-month intervals, requiring a face-to-face clinician visit. Wireless care involved more frequent monitoring and intervention in the event of anomalies in treatment use or effectiveness.

DETAILED DESCRIPTION:
Prior to enrollment, patients were seen by a clinician at the Veterans Administration (VA) Hospital in West Haven, Connecticut. Either a facility-based diagnostic polysomnogram or unattended home sleep testing was performed at the evaluating clinician's discretion. Clinicians that saw the patient determined whether PAP therapy was needed, and either auto-titrating continuous positive airway pressure (CPAP) or set pressures of CPAP were ordered for the patient. Patients received education about OSA and about their equipment from a respiratory therapist and physician's assistant within the VA who then provided the equipment for them. Patients coming to this internal Durable Medical Equipment (DME) provider were screened for participation in the study.The study was overseen by the Institutional Review Board at the Veterans Affairs Connecticut Health Care in West Haven, Connecticut. Informed consent was obtained from all participants.

Patients were included in the study if they were diagnosed with OSA (defined as AHI or apnea-hypopnea index greater than five per hour with symptoms, or AHI greater than 15/hour), and if they were being exposed to PAP for the first time. Patients who were previously treated with PAP, had central apnea, chronic respiratory failure, recent in-patient hospital admissions (=< 2 weeks), or were living outside cellular network coverage area were excluded from the study.

Patients that met study inclusion criteria were provided ResMed S9 devices with wireless modems. Their usage and treatment data was tracked using EasyCare Online, a cloud-based system for the ResMed devices. After the initial setup and educational settings, the patients received supplies as needed and troubleshooting of side effects of treatment as needed. Devices were not removed after 3 months if they were not adherent.

Patients in the usual care group were monitored on a 3-month, 6-month, 9-month and 12-month intervals with scheduling face-to-face visits. Adherence and efficacy data were only assessed by the clinician at these intervals.

Patients in the wireless care group were monitored more frequently using wireless modems as the method to obtain adherence and efficacy data.

We then determined adherence using CMS (Centers for Medicare & Medicaid Services) criteria at 3 months, and at 12 months. To obtain this data, we evaluated whether the PAP devices were used for 4 or more hours per night on 70% of nights during a consecutive 30-day period anytime during the first 3 months of initial use, and then a consecutive 30-day period in months 4-12. We also examined the daily use from the first to last day looking of overall patterns of utilization monthly, quarterly, semiannually and annually. Data was collected and maintained in a REDCap database (REDCap is a secure web application for building and managing online surveys and databases). Sensitivity and specificity calculations were then performed to evaluate predictability of adherence at 1 year using adherence at 3 months. Fisher's exact test was also used to evaluate the association between adherence at 3 months and 1 year and the association between AHI (Apnea -Hypopnea Index) and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed OSA patients
* AHI of 5/hour or greater
* Prescribed CPAP therapy
* Able to comply with treatment and understand treatment instructions

Exclusion Criteria:

* Not able to understand study requirements
* Significant cardiorespiratory disease - e.g. COPD (chronic obstructive pulmonary disease), severe CHF (congestive heart failure)
* Clinical instability at time of apnea diagnosis
* Prescribed BiPap (bilevel positive airway pressure) or ASV (Adaptive Support Ventilation), which are other types of PAP

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meir Kryger, MD, Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Health System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Naik S, Al-Halawani M, Kreinin I, Kryger M. Centers for Medicare and Medicaid Services Positive Airway Pressure Adherence Criteria May Limit Treatment to Many Medicare Beneficiaries. J Clin Sleep Med. 2019 Feb 15;15(2):245-251. doi: 10.5664/jcsm.7626. PMID 30736874

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: These patients will be monitored on a 3-month, 6-month, 9-month and 12-month intervals with face-to-face visits. Adherence and efficacy data will only be assessed by the clinician at these intervals.
  Monitoring every 3 months by face-to-face visits
- Wireless Care: These patients will be monitored using wireless modems as the method to obtain adherence and efficacy data.
  Frequent remote monitoring
Period: Overall Study
Arm/Group | Usual Care | Wireless Care
Started | 26 | 26
Completed | 22 | 20
Not Completed | 4 | 6
Not completed — Physician Decision | 4 | 4
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Wireless Care | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 22 | 36
  >=65 years | 12 | 4 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 21 | 24 | 45
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 3 | 5 | 8
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Airway Pressure Treatment Adherence in the First 3 Months
Description: Positive Airway Pressure Treatment Adherence defined as mean PAP use being > 4 hours per night for greater than 70% of nights.
Time Frame: First 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Wireless Care
Number analyzed (Participants) | 22 | 20
Participants | 10 | 9
Statistical Analysis 1: Comparison: Usual Care vs Wireless Care; PAP devices delivery to the patients was outsourced by the institution eliminating the point of recruitment for the study at our department. The recruitment was halted and the study proceeded with the follow-up of already recruited patients. As a result of the limited recruitment, planned statistical data analysis was not performed on the primary outcomes due to the smaller then expected number of subjects (expected 110 subjects in the Usual arm and 110 subjects in the Wireless arm; Test type: Other — Exact Fisher test was used on the collected information from the limited population; p < 0.01, Fisher Exact — Hypothesis: Active continuous monitoring of PAP treatment in OSA will result in improved adherence at 90 days Exact Fisher test was used on the collected information from the limited population; Exact Fisher test was used on the information from the limited population; Fisher exact test statistic value = 1; Exact Fisher test was used on the collected information from the limited population

2. Primary Outcome: Number of Participants With Positive Airway Pressure Treatment Adherence After 3 Months
Description: Demonstrated Periodic Adherence After 3 Months of Treatment During 4-12 months defined as mean PAP use being > 4 hours per night for greater than 70% of nights
Time Frame: 4-12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Wireless Care
Number analyzed (Participants) | 22 | 20
Participants | 10 | 10
Statistical Analysis 1: Comparison: Usual Care vs Wireless Care; CPAP devices delivery to the patients was outsourced by the institution eliminating the point of recruitment for the study at our department The recruitment was halted and the study proceeded with the follow-up of already recruited patients. As a result of the limited recruitment, planned statistical data analysis was not performed on the primary outcomes due to the smaller then expected number of subjects (expected 110 subjects in the Usual arm and 110 subjects in the Wireless arm; Test type: Other — Exact Fisher test was used on the collected information from the limited population; p < 0.01, Fisher Exact — Hypothesis: Active continuous monitoring of PAP treatment in OSA (Wireless group) will result in improved adherence at 90 days compared to Usual Group. Exact Fisher test was used on the collected information from the limited population; Exact Fisher test was used on the information from the limited population; Fisher exact test statistic value = 1; Exact Fisher test was used on the collected information from the limited population

3. Secondary Outcome: Receiving Effective Treatment for Obstructive Sleep Apnea
Description: Evaluate whether patients are effectively being treated with PAP or with alternate means of treatment for OSA (obstructive sleep apnea) at the end of 12 months.
Time Frame: 12 months
Population: 1 subject from the Wireless group was assigned to Provent treatment. 1 subject from the Usual group was assigned to Dental device treatment. Both subjects stopped using PAP and PAP monitoring and were considered not receiving effective PAP treatment for obstructive sleep apnea. Both subjects were lost in follow-up for our research study.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Wireless Care
Number analyzed (Participants) | 22 | 20
Participants | 10 | 10
Statistical Analysis 1: Comparison: Usual Care vs Wireless Care; [analysis description as in outcome 2, analysis 1]; Test type: Other — Exact Fisher test was used on the collected information from the limited population; p < 0.01, Fisher Exact — Hypothesis - Number of patients effectively treated with the PAP will be higher in the Wireless Group compared to the Usual Group Exact Fisher test was used on the collected information from the limited population; Estimation Parameter Other[Fisher exact = 1

4. Post Hoc Outcome: PAP Treatment Adherence in the First 3 Months of Treatment Compared to the PAP Treatment Adherence in the Next 9 Months of Treatment
Description: PAP treatment Adherence in the first 3 months of treatment (according to the CMS - Centers for Medicare & Medicaid Services - criteria) was compared to the PAP treatment Adherence in the next 9 months of treatment to verify the predictability of initial adherence or non-adherence for the future adherence or non-adherence (during the year) to PAP treatment. Adherence/non-adherence was analyzed based on the PAP usage reports (downloads) from the supplied PAP device, based on the yearly, quarterly and monthly portions of the reports.
  Patient data representing initial adherence or non-adherence and adherence or non-adherence during the year to PAP treatment was collected across both Usual care and Wireless Care Arms.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Initially Adherent Subjects: Subjects who became Adherent to the PAP treatment according to the CMS criteria within the first 3 months of treatment
- Initially Non-Adherent Subjects: Subjects who remained Non-Adherent to the PAP treatment according to the CMS criteria within the first 3 months of treatment
Arm/Group | Initially Adherent Subjects | Initially Non-Adherent Subjects
Number analyzed (Participants) | 19 | 23
Participants
  Adherent in the next 9 months | 13 | 7
  Non-Adherent in the next 9 months | 6 | 16
Statistical Analysis 1: Comparison: Initially Adherent Subjects vs Initially Non-Adherent Subjects; Exact Fisher test was used on the collected information from the limited population; Test type: Other — Exact Fisher test was used on the collected information from the limited population; p < 0.01, Fisher Exact — Hypothesis - PAP treatment Adherence in the first 3 months of treatment predicts the PAP treatment Adherence in the next 9 months of treatment Exact Fisher test was used on the collected information from the limited population; Other[Fisher exact test statistic value] = 0.0286 — Exact Fisher test was used on the collected information from the limited population; Exact Fisher test was used on the collected information from the limited population

5. Post Hoc Outcome: Adherence and AHI
Description: PAP adherence in subjects who had more than 20 respiratory events per hour during the initial sleep study was compared with the PAP adherence in subjects who had less than 20 respiratory events per hour during the initial sleep study.Patient data representing subjects who had more than 20 respiratory events per hour during the initial sleep study and subjects who had less than 20 respiratory events per hour during the initial sleep study was collected across both Usual care and Wireless Care Arms.
Time Frame: 1 year/12 months
Measure: Count of Participants; unit: Participants
Groups:
- AHI More Than 20: subjects who had more than 20 respiratory events per hour during the initial sleep study
- AHI Less Than 20: subjects who had less than 20 respiratory events per hour during the initial sleep study
Arm/Group | AHI More Than 20 | AHI Less Than 20
Number analyzed (Participants) | 23 | 19
Participants
  Adherent in 12 months | 19 | 7
  ANon-Adherent in 12 months | 4 | 12
Statistical Analysis 1: Comparison: AHI More Than 20 vs AHI Less Than 20; Exact Fisher test was used on the collected information from the limited population; Test type: Other — Exact Fisher test was used on the collected information from the limited population; p < 0.01, Fisher Exact — Hypothesis: Patients with the higher AHI are more likely to become adherent to the PAP therapy. Exact Fisher test was used on the collected information from the limited population; Exact Fisher test was used on the collected information from the limited population; Exact Fisher test = 0.0039; Exact Fisher test was used on the collected information from the limited population

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of time of subjects' participation in the study - 1 year or until a subject was withdrawn or terminated from the study
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, does not differ from the clinicaltrials.gov Definitions.
  Data was collected during the subject's follow-up and from the medical chart review.
Arm/Group | Usual Care | Wireless Care
All-Cause Mortality (participants affected / at risk) | 0/26 | 1/26
Serious Adverse Events (participants affected / at risk) | 3/26 | 3/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=26) | Wireless Care (N=26)
Acute Inpatient Psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Patient has long history of depression and anxiety. Patient stated his anxiety and depression has increased. Pt. Not suicidal, no hallucinations. Discharged in 3 days.Has outpatient psychiatric services.
Wolf -Parkinson-White syndrome. Hospitalization (Cardiac disorders) | 1 (1) | 0 (0) — Patient with WPW syndrome (Wolff-Parkinson-White syndrome) and previous ablation was hospitalized for sotabol load and discharged from to home in 3 days after achieving the goals of hospitalization with no restriction to physical activity
Hospitalisation due to Dyspnea and Chest Pain on exertion (Cardiac disorders) | 1 (1) | 0 (0) — A patient with a history of Myocardial Infarction presented with Dyspnea and Chest Pain on exertion. Troponins negative. Underwent nuclear stress test showed normal myocardial perfusion. Discharged home in 3 days
Hospitalization of encephalopathic patient transitioned to comfort care (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Participant with underlying cirrhosis of the liver, lung mass (possible cancer) and hepatocellular carcinoma was taken to a local civilian hospital. He was profoundly encephalopathic and transitioned to comfort care. Reported in mortality section.
Hospitalization Elective Laparoscopic repair of incisional hernia (Surgical and medical procedures) | 1 (1) | 0 (0) — Laparoscopic repair of incisional hernia complicated by post op ileus. Discharged in 9 days with scheduled follow up
Hospitalization for Elective Laminectomy - Fusion (Surgical and medical procedures) | 0 (0) | 1 (1) — Hospitalization for Elective Laminectomy - Fusion

LIMITATIONS AND CAVEATS:
CPAP was outsourced eliminating the point of recruitment which halted limiting the study proceeded to the follow-up of recruited patients. Planned statistical data analysis was not performed due to the smaller then expected numbers (expected 220)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes